CLINICAL TRIAL: NCT02914821
Title: Do Taxes Reduce the Purchasing of Soda?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Harvard University dining workers went on strike, we hope to relaunch in Fall 2017.
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Leslie John, Principal Investigator, Harvard University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB16-1285
Record Dates: First submitted 2016-09-03; First posted 2016-09-26 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Obesity; Diabetes
Keywords: consumption; decision making; policy; sweetened beverages; taxes; Diet, Food, and Nutrition
MeSH Terms: conditions — Obesity; Diabetes Mellitus

ARMS (4):
- Business as Usual (No "Tax") (No Intervention): Baseline data where business 'as usual' will be conducted and no price increases will be implemented on SSBs.
- General "Tax" (without named beneficiary) (Experimental): In the general tax condition investigators will introduce a 3 cent/ounce tax on the five SSB flavors the café offers. An example of this sign would be 'Pepsi, $2.29, includes 60 cent sugary drink surcharge.'
  Interventions: Behavioral: Simulated tax via 3 cent per ounce price increase
- Pre-K "Tax" (Experimental): In the Pre-K tax condition investigators will institute a 3 cent/ounce tax but will label the tax as proceeds going to Pre-K education. An example of this sign is, "Pepsi, $2.29, includes a 60 cent sugary drink surcharge to fund Pre-K education."
  Interventions: Behavioral: Simulated tax via 3 cent per ounce price increase
- Childhood Healthy Eating "Tax" (Experimental): In the Childhood Healthy Eating tax condition investigators will institute a 3 cent/ounce tax but will label the tax as proceeds going to Pre-K education. An example of this sign is, "Pepsi, $2.29, includes a 60 cent sugary drink surcharge to fund Childhood Healthy Eating education."
  Interventions: Behavioral: Simulated tax via 3 cent per ounce price increase

INTERVENTIONS:
Behavioral: Simulated tax via 3 cent per ounce price increase — For each of the 3 experimental conditions, investigators will increase the price of sugar-sweetened beverages by 3 cents per ounce. This price increase will be reflected in the price tag and described as a surcharge. In two of the arms (Pre-K and Childhood Healthy Eating), the beneficiary of the surcharge will be named.
  Arms: Childhood Healthy Eating "Tax"; General "Tax" (without named beneficiary); Pre-K "Tax"

SUMMARY:
The study will take place at a cafe managed by university dining services and is located in a university building adjacent to the psychology building. The cafe sells sugar-sweetened beverages and a variety of diet drinks. The campus dining services and the manager of the cafe have given investigators permission to "tax" their sugar sweetened beverages and will provide their sales data for a 12 week period.

The investigators will introduce four arms to the experiment. One arm will be baseline data where business 'as usual' will be conducted and no price increases will be implemented on SSBs. In the general tax condition the investigators will introduce a 3 cent/ounce tax on the five SSB flavors the café offers. In the Pre-K tax condition the investigators will institute a 3 cent/ounce tax but will label the tax as proceeds going to Pre-K education. This is designed after the Philadelphia tax that was recently passed where funds were earmarked to benefit childhood education. In the childhood healthy eating program condition the investigators will institute a 3 cent/ounce tax but will label the tax as proceeds going toward childhood healthy eating programs. In all tax conditions the firm will keep the proceeds, but the research team will make a donation to a Pre-K education non-profit and a childhood healthy eating non-profit of the amount generated by the tax during the study period.

Each experimental arm will run for 3 weeks total (for a total study period of 12 weeks). The conditions will alternate by week (i.e., week 1: business as usual; week 2: general tax; week 3: pre-K tax; week 4: childhood healthy eating tax; week 5: business as usual, etc). A research assistant will visit the café each week to make any necessary changes to signs that will label the drinks.

The investigators will change the signage of the drinks in the cooler during the study period. For the baseline period there will be no changes to the signs made. Currently all beverages are labeled with their name and cost (e.g., Pepsi, $1.89). In the tax conditions the investigators will change the price of the drink (3 cents/ounce) and add a line notifying consumers of the soda 'surcharge' (note "surcharge" will be used in the study because no tax was actually passed by the local government). An example of this sign would be 'Pepsi, $2.29, includes 40 cent sugary drink surcharge.' In the Pre-K tax condition an added line will say, "Pepsi, $2.29, includes a 40 cent sugar sweetened beverage surcharge. Proceeds benefit Pre-K education." In the childhood healthy eating programs condition the text will say, "Pepsi, $2.29, includes a 40 cent sugary drink surcharge. Proceeds benefit Childhood Healthy Eating programs."

DETAILED DESCRIPTION:
Diet-related diseases, such as diabetes and obesity, have become pervasive global health challenges, so much so that they are being called epidemics. The problem is particularly acute in the United States where two-thirds of adults and one-third of children are overweight or obese. A key contributor to increased dietary intake is the increased consumption of sugar-sweetened beverages.

Sugar-sweetened beverages (SSBs), also known as soft drinks, are beverages that are sweetened with sugar, high fructose corn syrup, or any other caloric sweetener; this excludes noncaloric (diet) drinks. The average American consumes approximately 47 gallons of SSBs per year. Americans consume about 278 calories more each day than they did 30 years ago and nearly half of this increase is attributable to increased consumption of SSBs. The consumption of SSBs has been cited as a key contributor to obesity and has been linked to other negative health problems, such as diabetes, heart disease, and dental cavities. Therefore, the increase in SSB consumption and the concurrent increase in diet-related diseases pose significant direct and indirect costs to society.

In response to these problems, health experts, laypeople and legislators alike advocate policies to reduce the consumption of SSBs. Several municipalities and states have proposed policies such as taxes, warning labels, and calorie labeling and a few have passed such policies. For example, Berkeley, CA recently adopted a SSB excise tax which charges an additional cent for each ounce of SSB sold. In June 2016, Philadelphia passed a 1.5 cent per ounce tax on sugary drinks and diet sodas.

The investigators believe it is critical to further test the effectiveness of taxes in the field. In this study, the investigators conduct a field experiment that tests different framing of taxes, namely whether the money is earmarked for a particular cause.

ELIGIBILITY:
Inclusion Criteria:

* All patrons who purchase a beverage at our study site (retail cafe) during the intervention are eligible for inclusion. The cafe is open to the public, though it primarily serves staff, patients and guests of the research labs in the building.

Exclusion Criteria:

* There are no exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Sugar-Sweetened Beverages Sold by Universal Product Code (UPC) | 3-week condition blocks
  Using the Universal Product Code (UPC) obtained in sales data, we will sum the total number of sugar sweetened beverages sold in each condition and can calculate this as a share of total beverages sold.

SECONDARY OUTCOMES:
Average Number of Beverage Calories Purchased Per Customer | 3-week condition blocks
  Using the UPCs and nutrition labels, we will calculate the average number of calories purchased that come from beverages.
Unsweetened Beverages Sold by Universal Product Code (UPC) | 3-week condition blocks
  Using the Universal Product Code (UPC) obtained in sales data, we will sum the total number of unsweetened beverages sold in each condition and can calculate this as a share of total beverages sold.
Changes in types of beverages purchased | 3 week condition blocks
  We will examine any changes in the types of beverages purchased during each condition, using the Universal Product Code (UPC) for bottled beverages. For example, if sugar-sweetened beverages sales decrease, do purchases of water increase?

IPD SHARING:
Plan to Share IPD: No